CLINICAL TRIAL: NCT02933775
Title: Autologous T Cells With a Chimeric Antigen Receptor in Patients With CD19-positive Malignant B Cell Leukemia and Lymphoma
Brief Title: CD19-redirected Autologous Cells (CAR-CD19 T Cells)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG3001
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: CD19 Positive Malignant B-cell Leukemia and Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR-CD19 T cells (Experimental): Autologous T Cells with a CD19-redirected Chimeric Antigen Receptor. Route of administration: Intravenous injection. Lymphodepleting conditioning regimen: A combination of fludarabine and cyclophosphamide will be administered at Day -9 - Day -4.
  Interventions: Genetic: CAR-CD19 T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: CAR-CD19 T cells — Initial dose: A total of 1 - 10×10^7 CAR-CD19 T cells/kg will be administered by 1 - 3 infusions. Subsequent dose will be based on the subject's response to initial dose.
  Other Names: CD19 Redirected Autologous Cells
Drug: Fludarabine — 30 mg/m^2/day×4 days
Drug: Cyclophosphamide — 500 mg/m^2/day×2 days

SUMMARY:
This study is designed for determining the safety and relative engraftment levels of the redirected autologous T cells transduced with the anti-CD19 lentiviral vector in patients with CD19-positive B cell leukemia and malignant lymphoma.

DETAILED DESCRIPTION:
A single arm open-label pilot study is designed to determine the safety, tolerability and engraftment potential of CAR-CD19 T cells in patients with CD19-positive malignant B cell leukemia and lymphoma. All subjects will receive CAR-CD19 T cells infusion.

Primary objectives:

1. Determine the safety and feasibility of the chimeric antigen receptor T cells transduced with the anti-CD19 lentiviral vector (referred to as "CAR-CD19 T" cells).
2. Determine the duration of in vivo survival of CAR-CD19 T cells.

Secondary objectives:

1. For patients with detectable disease, measure anti-tumor response due to CAR-CD19 T cells infusions.
2. To determine the amplification and survival of CAR-CD19 T 4-1BB:CD3ζ and CD28:CD3ζ as measured by the relative engraftment levels of CAR-CD19 T 4-1BB:CD3ζ and CD28:CD3ζ cells over time.
3. Estimate relative trafficking of CAR-CD19 T cells to tumors in bone marrow and lymphnodes.
4. Determine if cellular or humoral host immunity develops against the murine anti-CD19, and assess correlation with loss of detectable CAR-CD19 T (loss of engraftment).
5. Determine the relative subsets of CAR-CD19 T cells.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented CD19-positive malignant B cell leukemia and lymphoma.

  1. Patients aged between 18 ~ 65 with malignant B cell leukemia and lymphoma.
  2. CD19-positive B cell leukemia or lymphoma.
  3. Expected survival > 12 weeks.
  4. ECOG scores 0-1, or KPS scores > 80.
  5. Adequate venous access for apheresis or venous sampling, and no other contraindications for leukapheresis.
  6. WBC ≥ 2.5×109/L; LY ≥ 0.7×109/L; LY% ≥ 15%.
  7. Creatinine ≤ 2.0 mg/dL (176.8 μmol/L).
  8. ALT/AST ≤ 2.5 ULN.
  9. Bilirubin ≤ 2.0 mg/dL (34.2 μmol/L).
  10. Prothrombin Time (PT) : International Normalized Ratio (INR) < 1.7, or PT is at most 4 s longer than normal value.

All tests results should comply with the above criteria. No continuing supportive care is received.

Exclusion Criteria:

* 1. CD19-negative B cell leukemia or lymphoma. 2. Feasibility assessment during screening demonstrates < 5% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to αCD3/CD28 costimulation.

  3. Pregnant or lactating women. (The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion.) 4. Active hepatitis B or hepatitis C infection. 5. HIV/AIDS infection. 6. Uncontrolled active infection. 7. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.

  8. Previously treatment with any gene therapy products. 9. Allergy to immunotherapy and associated drugs. 10. Patients with heart disease that is in need of treatment or with poorly controlled hypertension determined by investigators.

  11. Patients with unstable or active ulceration or with gastrointestinal bleeding.

  12. Patients with previous or planed organ transplantation. 13. Hyponatremia with concentration of sodium in the blood < 125 mmol/L. 14. Serum potassium (baseline) < 3.5 mmol/L (Patients can take potassium supplements to recover serum potassium level prior to participating the study).

  15. Patients need anticoagulant (e.g. Warfarin or heparin). 16. Patients need long-term antiplatelet agent (Aspirin, dose > 300 mg/d; Clopidogrel, dose > 75 mg/d).

  17. Any radiotherapy conducted within 4 weeks prior to blood sampling.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-04 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Study related adverse events | 24 weeks
  Occurrence of study related adverse events, defined as NCI CTC ≥ Grade 3 signs/symptoms, laboratory toxicities and clinical events that are possible, likely or definitely related to study treatment at any time from the infusion until week 24, including infusional toxicity and any toxicity possibly related to the CAR-CD19 T cells.

SECONDARY OUTCOMES:
Primary engraftment endpoint | 2 years
  Duration of in vivo survival of CAR-CD19 T cells is defined as "engraftment". The primary engraftment endpoint is the # DNA vector copies per mg blood of CAR-CD19 T cells on week 4 after the first infusion. Q-PCR for CAR-CD19 T vector sequences will also be performed after infusion at 24 hours, weekly x 4, monthly x 6, and every 3 months thereafter until any 2 sequential tests are negative documenting loss of CAR-CD19 T cells.
Anti-tumor responses | 2 years
  Describe anti-tumor responses to CAR-CD19 T cell infusions.
Overall survival | 2 years
  Describe overall survival and cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Fangyuan Chen, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338